CLINICAL TRIAL: NCT05701267
Title: Neuro MRI Biomarkers for Treatment Navigation in Depression
Acronym: NEUROTREND
Status: Completed | Type: Observational
Sponsor: Eindhoven University of Technology (Other)
Collaborators: Clinical Trial Center Maastricht B.V. (Other)
Responsible Party: Sponsor
Other Study IDs: Neurotrend_001
Record Dates: First submitted 2022-02-22; First posted 2023-01-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MDD: Major depressive disorder patients (unipolar)
  Interventions: Device: MRI research
- CON: (Control) non-depressed
  Interventions: Device: MRI research

INTERVENTIONS:
Device: MRI research — 3T MRI protocol of ~1 hour

SUMMARY:
Background of the study:

Major depressive disorder is a severe neuropsychiatric condition that affects approximately 15% to 18% of people worldwide during their lifetime (Malhi & Mann, 2018). Selection of the optimal treatment is difficult.

A certain correlation (functional / structural, vascular or a mix of both) is expected between clinical data (obtained from psychometric tests such as the HDRS and psychiatric evaluations) and MRI parameters (functional activity, structural connectivity, anatomical variations, perfusion / diffusion etc.).

Objective of the study:

Identification of MRI-based biomarkers to predict clinical outcome of major depressive disorder in comparison with healthy controls. Outcome is defined by level of depressive and cognitive symptomatology and related comorbidity.

Study design:

An independent treating physician will inform a potentially eligible patient and ask whether he/she is interested in voluntary participation in the study. If he/she is interested, the independent treating physician will refer the patient to one of the clinicians from the GGz who is also involved in the Neurotrend study for further steps such as providing the information letter / informed consent and scheduling an intake interview at least one week after receiving all necessary information. Healthy controls will be recruited through public advertisement and via the website www.neurotrend.nl. Pilot subjects will be recruited from the Eindhoven University community and via the website www.neurotrend.nl. Both groups, healthy controls and pilot subjects, will have at least one week to consider and decide on participation. One week later an intake session will take place in which the inclusion and exclusion criteria will be checked. During this session, patients can also ask questions about the study and the informed consent will be signed if the participant is willing to participate voluntarily in the study. Subsequently at the end of the intake session, a starting (baseline) date will be planned for this participant . The actual participation starts at baseline. In total, 120 depressed patients and 60 healthy controls will participate in the study.

Each participant visits Kempenhaeghe twice, whereby each session, is dedicated to complete questionnaires and cognitive tests, such as memory tasks and eye tracking. In the last hour, the participant will be scanned (MRI). Two weeks before each visit, the participant has to fill in some questionnaires that have been sent to the participant.

Study population:

120 patients with major depressive disorder and 60 healthy controls*.

* Inclusion of up to 30 healthy "pilot" participants for technical evaluation. See above.

Primary study parameters/outcome of the study:

* Hamilton Depression Rating Scale (HDRS) scores
* Treatment / medication usage
* MRI metrics (varies per MRI modality, an example is volume per region for a T1-weighted scan and fractional anisotropy for diffusion-weighted scans).

Secondary study parameters/outcome of the study (if applicable):

* Scores of psychometric assessments (e.g. STAI-DY1 - anxiety score)
* Scores of cognitive assessments (e.g. average response time for the eye-tracking task)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

The participant burden is low and is divided into an intake session and two research sessions. The MRI scan is non-invasive, and subjects can indicate that they want to stop the scan at any time during the scan by squeezing a type of balloon that will lie next to the subject in the case that they feel uncomfortable or for any other reason. Subjects with MRI contraindications (e.g.

claustrophobia, pregnancy or implants not suitable for MRI) are already excluded in advance and will therefore not participate in the study at all. Mostly, the subjects will lie still during the scan, except for one affective task in which they will be asked to match different emotional faces for about 5 minutes.The cognitive tests will only consist of memory, reaction speed, attention, and processing speed tasks which in total, do not last more than 30 minutes. The risks of the MRI scanner (CE-marked) are minimal.

DETAILED DESCRIPTION:
Limitation to research to date

Heterogeneous findings of current studies may indicate that MDD has been approached too much as a homogeneous concept, whereas analysing subtypes might be more useful. The literature supports the existence of different MDD subtypes based on biological variables and/or clinical features. Research has distinguished 3 types of MDD based on depressive, symptomatology: a severe melancholic class, a severe atypical class and a class of moderate severity. Both depression severity (moderate vs severe) and the nature of depressive symptoms (melancholic vs atypical) were found to be important differentiators between those subtypes. Other subgroups of relevance may be remission vs. non-remission, early onset vs. late onset depression. The relation with neuroimaging findings is scarce and inconsistent. As depressive symptoms may also strongly fluctuate over time, repeated MRI and clinical data acquisition at different points in time is warranted. There is a relative scarcity of longitudinal MRI studies on MDD. Large representative samples are warranted, addressing multiple factors such as sociodemographic characteristics, clinical history (incl. childhood trauma), co-morbidity and monitoring of treatment, including type and duration. This will elucidate causative mechanisms as well as the role of treatment, which may pave the path towards diagnostic subtyping and treatment navigation. Moreover, brain alterations are usually described on a structural, functional and vascular level and seldom from an integral approach, let alone in a longitudinal design. A multi-modal approach whereby the three levels are considered might thus increase the reproducibility of findings. In addition, there is an urgent need to find biomarkers that are meaningful on the individual patient level. Machine learning is a technique that can be utilized to allow imaging risk markers to be identified at the level of subtypes and ultimately on the individual level, which is crucial for clinical applicability.

Current study

The Neurotrend study will contribute to the existing literature by aiming to predict outcome in MDD using multi-modal imaging with an observational study design. Two scanning sessions with one year in between will be held for patients with MDD and controls, as well as a broad assessment of clinical, cognitive and demographic variables (at baseline and 1-year follow-up). Predicting outcome at the level of subtypes/individuals in a naturalistic clinical setting is a different approach to identify biomarkers than most studies have done so far. For this purpose, machine learning will be used, which is a powerful method to identify biomarkers from the different MRI modalities. For the first time, IVIM and T2*-weighted imaging will be included in the MRI protocol to yield more insight into the microvascularity and microbleeds of the brain. In addition, other novel techniques will be applied to increase the chance of finding meaningful biomarkers. For instance, with respect to the brain alterations on a structural level, high spatial resolutions (using multiband imaging) and better automated segmentation methods will be used to examine the substructures of brain regions with high accuracy as substructural imaging is becoming more popular and could identify more reliable biomarkers. For the brain alterations on a functional level, multiband and multi-echo imaging lead to higher spatial/temporal resolution which will help to reduce the noise and artifacts to which fMRI is very susceptible.

ELIGIBILITY:
MDD patients:

Inclusion Criteria:

Satisfy DSM-5 clinical criteria for MDD (acute and subacute duration)

* Unipolar depression (i.e. no bipolar depression/mania)
* Age: 18-65 (m/f)
* Willing and able to provide informed consent and agree that incidental findings are reported

Exclusion Criteria:

* Concurrent neurological disorder (e.g. epilepsy, stroke, head trauma, etc.)
* Current substance or alcohol abuse
* History of psychosis, bipolar depression, autism spectrum disorder, attention deficit hyperactivity disorder or (mild) intellectual disability
* Contra-indication for MRI (see MRI safety form), includes implants, tattoos non-compatible with brain MRI, pregnancy, claustrophobia) Previous or current treatment with electroconvulsive therapy (ECT), deep-brain stimulation (DBS) or transcranial magnetic stimulation (TMS)
* More than 3 depressive episodes in the past

  60 healthy controls

Inclusion Criteria:

* Age: 18-65 (m/f)
* Willing and able to provide informed consent and agree that incidental findings are reported

Exclusion Criteria:

* A neurological disorder (e.g. epilepsy, stroke, head trauma, etc.)
* Current substance or alcohol abuse
* History of psychosis, bipolar depression, autism spectrum disorder, attention deficit and hyperactivity disorder or (mild) intellectual disability
* Contra-indication for MRI (see MRI safety form), includes implants, tattoos non-compatible with brain MRI, pregnancy, claustrophobia)
* Has a current episode of a MDD or ever had an MDD
* Previous or current treatment with electroconvulsive therapy (ECT), deep-brain stimulation (DBS) or transcranial magnetic stimulation (TMS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MMD versus (controls) non-depressed
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Basline brain region (subfield) volumes | baseline
  Volumes are extracted from T1w and T2w scans. Subfield volumes of the hippocampus and amygdala can be extracted from a high-resolution T2w image.
1-Year brain region (subfield) volumes | 1 year
  Volumes are extracted from T1w and T2w scans. Subfield volumes of the hippocampus and amygdala can be extracted from a high-resolution T2w image.
Baseline microvascular pseudodiffusion | baseline
  Intravoxel incoherent motion assesses perfusion in the small vessels of the brain.
Baseline microvascular perfusion fraction | baseline
  Intravoxel incoherent motion assesses perfusion in the small vessels of the brain.
1-Year microvascular pseudodiffusion | 1 year
  Intravoxel incoherent motion assesses perfusion in the small vessels of the brain.
1-Year microvascular perfusion fraction | 1 year
  Intravoxel incoherent motion assesses perfusion in the small vessels of the brain.
Baseline white matter hyperintensity volumes | baseline
  The FLAIR scan attenuates the CSF signal and therefore, it is excellent in distinguishing white-matter abnormalities surrounding the CSF.
1-Year white matter hyperintensity volumes | 1 year
  The FLAIR scan attenuates the CSF signal and therefore, it is excellent in distinguishing white-matter abnormalities surrounding the CSF.
Baseline structural connectivity (DTI) fractional anisotropy | baseline
  This T2*-weighted scan will measure the anatomical connections between brain areas.
Baseline structural connectivity (DTI) vessel density | baseline
  This T2*-weighted scan will measure the anatomical connections between brain areas.
1-Year structural connectivity (DTI) fractional anisotropy | 1 year
  This T2*-weighted scan will measure the anatomical connections between brain areas.
1-Year structural connectivity (DTI) vessel density | 1 year
  This T2*-weighted scan will measure the anatomical connections between brain areas.
Baseline activity in regions involved in emotion processing | baseline
  Task-based fMRI will assess activity in, amongst others, the amygdala and anterior cingulate cortex. Activity is expressed in t-values between activity (average measured BOLD signal in region-of-interest) in two conditions/contrasts:
  Faces versus Rest Faces versus Shapes
1-Year activity in regions involved in emotion processing | 1 year
  Task-based fMRI will assess activity in, amongst others, the amygdala and anterior cingulate cortex. Activity is expressed in t-values between activity (average measured BOLD signal in region-of-interest) in two conditions/contrasts:
  Faces versus Rest Faces versus Shapes
Baseline functional connectivity and derivatives thereof | baseline
  Resting-state fMRI will assess functional connectivity between brain regions and networks. Derivations include e.g. directed or time varying functional connectivity.
1-Year functional connectivity and derivatives thereof | 1 year
  Resting-state fMRI will assess functional connectivity between brain regions and networks. Derivations include e.g. directed or time varying functional connectivity.
Baseline cerebral blood flow | baseline
  Arterial spin labeling measures blood flow from which cerebral blood flow can be extracted
1-Year cerebral blood flow | 1 year
  Arterial spin labeling measures blood flow from which cerebral blood flow can be extracted
Baseline total volume microbleeds (susceptibility-weighted imaging) | baseline
  This T2*-weighted scan is used to detect brain microbleeds
Baseline total number of microbleeds (susceptibility-weighted imaging) | baseline
  This T2*-weighted scan is used to detect brain microbleeds
1-Year total volume microbleeds (susceptibility-weighted imaging) | 1 year
  This T2*-weighted scan is used to detect brain microbleeds
1-Year total number of microbleeds (susceptibility-weighted imaging) | 1 year
  This T2*-weighted scan is used to detect brain microbleeds
Baseline depression severity score | baseline
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.
3-Months depression severity score | 3 months
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.
6-Months depression severity score | 6 months
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.
9-Months depression severity score | 9 months
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.
1-Year depression severity score | 1 year
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.
Baseline depression severity score | At baseline
  Full spectrum of symptoms assessed via the Hamilton Depression Rating Scale (HDRS) 17 questionnaire. 17 items are rated from 0-4 or 0-2. Total scores ranges from 0-51. The HDRS includes questions regarding symptoms such as: depressed mood, feelings of guilt, suicide, anxiety and more.

SECONDARY OUTCOMES:
Sleep score | At baseline and after 1 year
  As assessed from the insomnia severity index questionnaire. 7 items are scored from 0-4. Range scores: 0-28. Higher score ---> More insomnia-related symptoms.
Anxiety score | At baseline and after 1 year
  As assessed from the State-Trait Anxiety Inventory Dutch Y 1 (STAI-DY1) questionnaire. 20 items are scored from 1-5. Range scores: 20-100. Higher score --> More anxiety-related symptoms
Neuroticism score | At baseline and after 1 year
  As assessed from the Neuroticism, Extraversion, Openness to Experiences Five-Factor Inventory (NEO-FFI) questionnaire. 60 items can be scored from 1-5. Range scores: 60-300. Higher scores ---> more symptoms related to neuroticism.
Childhood trauma score | At baseline and after 1 year
  As assessed from the Childhood trauma questionnaire (Dutch: JTV) - long version. 28 items can be scored from 1-5. Range scores: 28-140. Higher score --> More traumatic experience during childhood.
Psychosis score | At baseline and after 1 year
  As assessed from the Community Assessment of Psychic Experience (CAPE) questionnaire. 42 items range from 0-3. If an item is scored from 1-3, a more detailed question should be filled in ranging from 0-3. Range scores: 0-252 (42 * (3 * 2)). Higher scores --> more psychotic symptoms.
Comorbidities | At baseline and after 1 year
  As assessed from the MINI neuropsychiatric interview. No scores/scale. Labels indicate different comorbidities that might be crucial for biological subtype identification.
Medication and treatment | Every 3 months for MDD - At baseline and 1 year follow-up for healthy controls
  Custom questionnaire to assess type and dose of medication and types of treatments received. No scores and no scale.
Psychomotor speed and reaction time | At baseline and after 1 year
  As assessed by an eye-tracker camera and custom task in Tobii software Subjects have to focus on a white block appearing multiple times on a black background. It is an indication of medication influence on cognition. No scale; faster reaction times indicate higher performance.
Attention and processing speed | At baseline and after 1 year
  As assessed by FEPSY software. Includes visual reaction times and pattern recognition tasks. No scale; faster reaction times indicate higher performance.
Long and short-term verbal memory | At baseline and after 1 year
  As assessed by the RVALT (15 words memory and recall test). Each repetition a score from 1-15 can be achieved; higher scores indicate higher performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Kempenhaeghe, Heeze, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
No plan available yet